CLINICAL TRIAL: NCT06740734
Title: The Effect of Stress Ball and Expressive Touch Application on Pain, Mobilization and Breastfeeding During Episiotomy Repair
Brief Title: The Effect of Stress Ball and Expressive Touch Application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mine Gokduman Keles (Other)
Responsible Party: Sponsor-Investigator, Mine Gokduman Keles, Asst.Prof. Mine GÖKDUMAN KELEŞ PhD. Midwifery Department, Burdur Mehmet Akif Ersoy University
Organization: Burdur Mehmet Akif Ersoy University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Burdur Mehmet Akif Ersoy Unive
Record Dates: First submitted 2024-12-06; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Birth Trauma
Keywords: Pain Management; Midwifery; Episiotomy; Stress Ball; Expressive Touch
MeSH Terms: conditions — Birth Injuries; Agnosia

STUDY DESIGN:
Intervention Model Description: Intervention The pregnant women who were randomly included in the study and control groups by going to the clinic during the study period by the researcher will first fill out the "Informed Volunteer Consent Form" and "Pregnant Identifier Form (Pregnant Identifier Information-Labor and Episiotomy Follow-up Form first 8 questions)".
  Implementation process
  * Group 1; Stress ball
  * Group 2 Expressive touch after cesarean
  * Control Group will be given routine care.
  Study Group 1: Sterile Stress ball during mediolateral episiotomy repair for pregnant women who received stress ball application. Participants in the stress ball group will be asked to squeeze and loosen the stress ball in their hand (Ozen et al., 2023).
  Group 3 -Those who received expressive touch During mediolateral episiotomy repair, expressive touch will be applied to one of the mother's hands by the researcher for an average of 15-20 minutes (Association, 2023.).
  In the Control Group The women in the control group receiv
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The group will be given routine care
- Stress ball (Active Comparator): Sterile Stress ball applied to pregnant women during mediolateral episiotomy repair. Participants in the stress ball group will be asked to squeeze and loosen the stress ball in their hands
  Interventions: Behavioral: Stress ball
- Expressive touch applications (Active Comparator): During the mediolateral episiotomy repair, expressive touch will be applied to one hand of the mother by the researcher, lasting approximately 15-20 minutes.
  Interventions: Behavioral: Expressive touch applications

INTERVENTIONS:
Behavioral: Stress ball — Sterile Stress ball for pregnant women during mediolateral episiotomy repair. Participants in the stress ball group will be asked to squeeze and loosen the stress ball in their hands.
  Arms: Stress ball
Behavioral: Expressive touch applications — During the mediolateral episiotomy repair, expressive touch will be applied to one hand of the mother by the researcher, lasting approximately 15-20 minutes
  Arms: Expressive touch applications

SUMMARY:
Purpose: The study will be conducted to examine the effects of stress ball and expressive touch application on pain, mobilization and breastfeeding during episiotomy repair. Materials and Methods: In the randomized controlled experimental study, data will be obtained using the "VAS pain score", "6 Minute Walk Test" Bristol Breastfeeding Assessment Scale. Stress Ball and Expressive Touch will be applied to the women in the study group during the episiotomy application and no application will be applied to the patients in the control group during the procedure.

DETAILED DESCRIPTION:
Introduction Episiotomy is a controlled surgical incision made in the perineum to widen the vaginal opening in the second stage of labor . Although limited and indicated use of episiotomy is recommended, it is applied in around 40%.

Episiotomy procedure is observed to affect sexual health in the short term; pain, anxiety, limited mobility, difficulties in micturition and defecation . In the long term, it is seen that the fear of episiotomy in pregnant women increases the rate of elective cesarean section . The use of sleep-inducing drugs to reduce pain during episiotomy repair can cause side effects such as changes in fetal heart rate and decrease in maternal blood pressure . Evidence-based practices recommend the use of various nonpharmacological methods to reduce pain during episiotomy repair . Evidence-based practices support stress ball and expressive touch in pain management .

Stress ball; is a nonpharmacological method that reduces the feeling of pain by pulling pain-related receptors in the brain to another point.In the literature, stress ball is seen to be used to reduce pain during endoscopy , peripheral intravenous catheter application ,, and gynecological procedures .Again, expressive Touch is an approach that aims to regulate, increase, balance and protect energy to heal diseases or symptoms caused by imbalance in vital energy fields .It is a consciously directed energy exchange in which the practitioner uses their hands as a focal point to facilitate the process .It has been reported in the literature that expressive touch reduces women's pain in labor .Women in labor and early postpartum need verbal and nonverbal communication from midwives .

Reducing pain during episiotomy repair is available in the literature .However, there are limited studies on long-term results .. In the current literature, it was aimed to determine the effects of stress ball and expressive touch application on pain, mobilization and breastfeeding during episiotomy repair and to pioneer future research. It is thought that the results obtained in this study will significantly contribute to women's positive birth experiences and the development of midwifery practices.

ELIGIBILITY:
Inclusion Criteria:

Women who speak Turkish, are between the ages of 18-35, primiparous, gestational age between 37-42, who have undergone mediolateral episiotomy,

-

Exclusion Criteria:

Women diagnosed with risky pregnancies, those with vision and hearing problems, those with deep lacerations during delivery, those with 3rd and 4th degree lacerations.

-

Ages: 18 Days to 35 Days | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — primiparous, pregnancy
Enrollment: 105 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 HOUR
  VAS pain score is used to evaluate pain severity. Pain on a numerical rating scale ranges from 0 (absence of pain) to 10 (unbearable pain).
Mobilization | 1 HOUR
  In the first 48 hours after birth, the first postpartum mobilization hour, duration, and the number of subsequent mobilizations will be recorded (Prokopowicz, Korzeniewska, Byrka, & Obstetrics, 2021). The decision to start or continue mobilization will be made by the healthcare professional working in the clinic.
  Women's mobilization status will be evaluated. The examiner will note the success or failure of the patient's mobilization along with its duration. (The beginning of the measurement was determined as the moment the patient got out of bed from a sitting position, and the end of the measurement was determined as the moment the patient returned to bed). If the patient got out of bed and started walking (took at least one step), he received a score of 1 (successful) on the questionnaire. If he stood up but did not take a single step while returning to a sitting position, he received a score of 0. Mobilization time was measured in minutes.
6-Minute Walk Test (6MWT) | 1 HOUR
  6MWT will be used to evaluate the physical functions of the patients. During this test, a 30-meter-long hard-surfaced track will be walked at a normal pace for six minutes. This track is marked every 3 meters and a cone is placed at the end of this 30-meter track and the same track is returned around it. The researcher will record the distance the patient walks in 6 minutes in meters. The test will be performed in a 60-meter long hospital corridor
Bristol Breastfeeding Assessment Scale; | 1 HOUR
  "Bristol Breastfeeding Assessment Scale (BEDÖ) was developed by Jenny Ingram in 2014 and adapted to Turkish by Dolgun and her friends in 2017 (İnal, Erdim, Korkut, & Dolgun). The scale was developed to evaluate breastfeeding problems and adequacy frequently encountered in the postpartum period. The mother is observed by a health professional during breastfeeding and the form is filled out by evaluating the mother and the baby in line with the criteria. The application time of the scale is 5-10 minutes. While the Cronbach's Alpha value of the original form of the tool was found to be 0.68, it was found to be 0.77 in the Turkish adaptation study. In our study, the reliability coefficient Chronbach's Alpha value was determined as ….. The measurement tool is a Likert-type scale consisting of 4 items: "positioning", "holding", "sucking" and "swallowing" (İnal et al.).

IPD SHARING:
Plan to Share IPD: No